CLINICAL TRIAL: NCT05771220
Title: Effectiveness of Radial Extracorporeal Shockwave Therapy Combined With Evidence-Based Physical Therapy for Adhesive Capsulitis Shoulder: A Randomized Controlled Trial
Brief Title: Radial Extracorporeal Shockwave Therapy Combined With Evidence-Based Physical Therapy for Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taif University (Other)
Responsible Party: Principal Investigator, Hosam Alzahrani, Assistant Professor; Department of Physical Therapy, Taif University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A01510
Record Dates: First submitted 2023-02-09; First posted 2023-03-16 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Adhesive Capsulitis of Shoulder
Keywords: Frozen shoulder; Extracorporeal shockwave therapy
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, single blinded, placebo
Who Masked: Participant
Masking Description: Single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- radial extracorporeal shockwave therapy+ evidence-based physical therapy (Experimental): radial extracorporeal shockwave therapy + evidence-based physical therapy
  Interventions: Other: radial extracorporeal shockwave therapy+ evidence-based physical therapy
- sham radial extracorporeal shockwave therapy + evidence-based physical therapy (Placebo Comparator): sham radial extracorporeal shockwave therapy+ evidence-based physical therapy
  Interventions: Other: sham radial extracorporeal shockwave therapy+ evidence-based physical therapy

INTERVENTIONS:
Other: radial extracorporeal shockwave therapy+ evidence-based physical therapy — The experimental group received six sessions of rESWT over six weeks in addition to an EBPT program. The rESWT procedure involved applying shockwaves to the affected area using a radial probe, with sessions lasting 10-15 minutes and consisting of up to 2000 impulses delivered at a frequency of 3-6 pulses per second and an energy intensity level of 1.8 bar, based on patient tolerance. Patients were seated or lying down during the rESWT procedure, with gel or oil applied to facilitate shockwave transmission through the skin. Additionally, participants received a 30-minute exercise program twice a week for 6 weeks, which included hot packs, stretching, range of motion exercises, and isometric shoulder and scapular exercises. They were also instructed to perform the same exercises at home daily.
  Arms: radial extracorporeal shockwave therapy+ evidence-based physical therapy
Other: sham radial extracorporeal shockwave therapy+ evidence-based physical therapy — The participants in the control group received six weeks of sham rESWT (radial extracorporeal shock wave therapy) combined with the EBPT (evidence-based physical therapy) program. The sham rESWT involved six sessions with a maximum of 200 impulses delivered at a low intensity, with the applicator placed on the affected area for the same duration as the experimental group. Additionally, participants received a 30-minute exercise program twice a week for 6 weeks, which included hot packs, stretching, range of motion exercises, and isometric shoulder and scapular exercises. They were also instructed to perform the same exercises at home daily.
  Arms: sham radial extracorporeal shockwave therapy + evidence-based physical therapy

SUMMARY:
The goal of this clinical trial is to evaluate the combined effects of radial extracorporeal shockwave therapy (rESWT) and evidence-based physical therapy (EBPT) interventions for patients with adhesive capsulitis. The main questions it aims to answer are:

What is the effectiveness of combining rESWT with EBPT interventions for the management of adhesive capsulitis compared to EBPT alone? How does the combination of rESWT and EBPT affect pain, range of motion, and functional outcomes in patients with adhesive capsulitis?

Researchers will compare rESWT plus EBPT to a sham rESWT plus EBPT to see if rESWT provides better results for subjects with adhesive capsulitis.

The study will randomly assign participants to receive either rESWT plus EBPT or sham rESWT plus EBPT over a 6-week intervention period. The primary outcomes will be pain and disability, while secondary outcomes will include shoulder range of motion, psychological distress, and health-related quality of life. These outcomes will be assessed at baseline, post-intervention, and 12 weeks post-randomization.

ELIGIBILITY:
Inclusion Criteria:

* Having a relapsed or episode of pain score ≥5 at the assessment with a past history of pain for at least 2 weeks.
* phase 1 or 2 frozen shoulder confirmed by a physician
* ROM restriction (>75% ROM loss in ≥2 directions including abduction, flexion and external rotation)
* no treatment other than analgesics with unresponsive ROM restriction for the past 2 months
* unwilling or waiting and did not undergo joint injection
* Diagnosed with shoulder adhesive capsulitis,
* ≥18 years
* Diabetes mellitus

Exclusion Criteria:

* bilateral shoulder involvement
* History of previous surgery on the shoulder
* Shoulder fracture
* Cancer
* Glenohumeral or Acromioclavicular arthritis
* Inflammatory disorders
* Bleeding disorders
* Presence of severe osteoporosis
* Pulmonary diseases
* Any neuromuscular disorders
* Pregnancy
* Implanted pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | baseline, and at 7 and 12 weeks
  Visual analogue scale for pain intensity measurement (0 (no pain) - 10 (worst pain))
Disabilities of the Arm, Shoulder, and Hand Quick version (DASH) | baseline, and at 7 and 12 weeks
  Shoulder disability was measured using the Disabilities of the Arm, Shoulder, and Hand Quick version (DASH) questionnaire (0-100). It's an 11-item questionnaire that measures a patient's ability to perform specific upper extremity tasks, and higher scores on the scale indicate a higher disability. The scale ranges from 0 to 100; where higher score indicates higher disability.

SECONDARY OUTCOMES:
Depression Anxiety Stress Scales (DASS-12) | baseline, and at 7 and 12 weeks
  Depression Anxiety Stress Scales, is made up of 12 self-report items. It is a 12-item self-report instrument designed to measure the three related negative emotional states of depression, anxiety, and tension/stress. It ranges 0-144, where higher score on the scale denotes higher endorsement of mental distress symptoms.
Short Form-12 | baseline, and at 7 and 12 weeks
  The 12-Item Short Form Health Survey questionnaire (SF-12; 0-100) is a very popular instrument for evaluating Health-Related Quality of Life.HIgher score on the scale indicates better Health-Related Quality of Life.
Range of Motion (passive and active) | baseline, and at 7 and 12 weeks
  Range of Motion is measured by goniometer. Higher score on goniometer indicates better range of motion.
  Flexion: 0-180 Abduction: 0-180 Internal rotation: 0-90 External rotation: 0-90

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Thager General Hospital, Jeddah, Mecca Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lee S, Lee S, Jeong M, Oh H, Lee K. The effects of extracorporeal shock wave therapy on pain and range of motion in patients with adhesive capsulitis. J Phys Ther Sci. 2017 Nov;29(11):1907-1909. doi: 10.1589/jpts.29.1907. Epub 2017 Nov 24. PMID 29200621
- [Result] Muthukrishnan R, Rashid AA, Al-Alkharji F. The effectiveness of extracorporeal shockwave therapy for frozen shoulder in patients with diabetes: randomized control trial. J Phys Ther Sci. 2019 Jul;31(7):493-497. doi: 10.1589/jpts.31.493. Epub 2019 Jul 2. PMID 31417208
- [Result] Kelley MJ, McClure PW, Leggin BG. Frozen shoulder: evidence and a proposed model guiding rehabilitation. J Orthop Sports Phys Ther. 2009 Feb;39(2):135-48. doi: 10.2519/jospt.2009.2916. PMID 19194024
- [Result] Vahdatpour B, Taheri P, Zade AZ, Moradian S. Efficacy of extracorporeal shockwave therapy in frozen shoulder. Int J Prev Med. 2014 Jul;5(7):875-81. PMID 25104999
- [Result] Le HV, Lee SJ, Nazarian A, Rodriguez EK. Adhesive capsulitis of the shoulder: review of pathophysiology and current clinical treatments. Shoulder Elbow. 2017 Apr;9(2):75-84. doi: 10.1177/1758573216676786. Epub 2016 Nov 7. PMID 28405218
- [Result] Cao DZ, Wang CL, Qing Z, Liu LD. Effectiveness of extracorporeal shock-wave therapy for frozen shoulder: A protocol for a systematic review of randomized controlled trial. Medicine (Baltimore). 2019 Feb;98(7):e14506. doi: 10.1097/MD.0000000000014506. PMID 30762780
- [Result] Nakandala P, Nanayakkara I, Wadugodapitiya S, Gawarammana I. The efficacy of physiotherapy interventions in the treatment of adhesive capsulitis: A systematic review. J Back Musculoskelet Rehabil. 2021;34(2):195-205. doi: 10.3233/BMR-200186. PMID 33185587
- [Result] Agarwal S, Raza S, Moiz JA, Anwer S, Alghadir AH. Effects of two different mobilization techniques on pain, range of motion and functional disability in patients with adhesive capsulitis: a comparative study. J Phys Ther Sci. 2016 Dec;28(12):3342-3349. doi: 10.1589/jpts.28.3342. Epub 2016 Dec 27. PMID 28174448
- [Result] Jain TK, Sharma NK. The effectiveness of physiotherapeutic interventions in treatment of frozen shoulder/adhesive capsulitis: a systematic review. J Back Musculoskelet Rehabil. 2014;27(3):247-73. doi: 10.3233/BMR-130443. PMID 24284277
- [Result] Yuan X, Zhou F, Zhang L, Zhang Z, Li J. Analgesic Effect of Extracorporeal Shock Wave Treatment Combined with Fascial Manipulation Theory for Adhesive Capsulitis of the Shoulder: A Retrospective Study. Biomed Res Int. 2018 Jan 18;2018:3450940. doi: 10.1155/2018/3450940. eCollection 2018. PMID 29581969
- [Result] Park C, Lee S, Yi CW, Lee K. The effects of extracorporeal shock wave therapy on frozen shoulder patients' pain and functions. J Phys Ther Sci. 2015 Dec;27(12):3659-61. doi: 10.1589/jpts.27.3659. Epub 2015 Dec 28. PMID 26834326
- [Result] Struyf F, Meeus M. Current evidence on physical therapy in patients with adhesive capsulitis: what are we missing? Clin Rheumatol. 2014 May;33(5):593-600. doi: 10.1007/s10067-013-2464-3. Epub 2013 Dec 28. PMID 24374758
- [Result] Zhang R, Wang Z, Liu R, Zhang N, Guo J, Huang Y. Extracorporeal Shockwave Therapy as an Adjunctive Therapy for Frozen Shoulder: A Systematic Review and Meta-analysis. Orthop J Sports Med. 2022 Feb 4;10(2):23259671211062222. doi: 10.1177/23259671211062222. eCollection 2022 Feb. PMID 35141337
- [Result] Qiao HY, Xin L, Wu SL. Analgesic effect of extracorporeal shock-wave therapy for frozen shoulder: A randomized controlled trial protocol. Medicine (Baltimore). 2020 Jul 31;99(31):e21399. doi: 10.1097/MD.0000000000021399. PMID 32756135
- [Derived] Sharahili TM, Alzahrani HA. Effect of radial extracorporeal shockwave therapy combined with evidence-based physical therapy for adhesive capsulitis of the shoulder: A randomized controlled trial. Saudi Med J. 2025 Jul;46(7):816-824. doi: 10.15537/smj.2025.46.7.20250213. PMID 40628437